CLINICAL TRIAL: NCT05789563
Title: Comparison of SpO2 Measurement Accuracy of Different Types of Smartwatches
Acronym: CSMADTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NVT_01_2023
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Hypoxia
Keywords: SpO2; Pulse oximetry; Smartwatch
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: All participants go through all study arms, in random order. Two measuring devices are active simultaneously during each measurement on each participant and their functioning is compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First smartwatch model (Experimental): Volunteers sequentially inhale three hypoxic gas mixtures each for 2.5 minute. Every measurement will begin with a two-minute stabilization phase, during which the physiological values of the volunteer will be checked. During the experiment, SpO2 measurements will be taken by hand from the watch and the pulse oximeter simultaneously.
  Interventions: Other: Hypoxia and Smartwatch model
- Second smartwatch model (Experimental): Volunteers sequentially inhale three hypoxic gas mixtures each for 2.5 minute. Every measurement will begin with a two-minute stabilization phase, during which the physiological values of the volunteer will be checked. During the experiment, SpO2 measurements will be taken by hand from the watch and the pulse oximeter simultaneously.
  Interventions: Other: Hypoxia and Smartwatch model
- Third smartwatch model (Experimental): Volunteers sequentially inhale three hypoxic gas mixtures each for 2.5 minute. Every measurement will begin with a two-minute stabilization phase, during which the physiological values of the volunteer will be checked. During the experiment, SpO2 measurements will be taken by hand from the watch and the pulse oximeter simultaneously.
  Interventions: Other: Hypoxia and Smartwatch model

INTERVENTIONS:
Other: Hypoxia and Smartwatch model — Breathing mixtures of O2 (14 %, 12 %, 10 %) balanced with N2 and monitoring SpO2 by one of the smartwatch models on left wrist and by pulse oximeter on left index finger.

SUMMARY:
The aim of the study is to compare the accuracy of peripheral blood oxygen saturation measurements using smartwatches from three manufacturers compared to a standard medical pulse oximeter.

DETAILED DESCRIPTION:
The aim is to create a study that compares multiple smartwatch models simultaneously with a standard medical pulse oximeter using a single measurement methodology. According to the available literature, no such study exists. The methodology of the study and the subsequent statistical evaluation are based on the guidelines of the standard ČSN EN ISO 80601-2-61, which specifies requirements for the basic safety and necessary functionality of pulse oximetry devices. The comparison will be performed non-invasively in healthy volunteers during gradual desaturation in the range of 70-100 % SpO2 (normobaric hypoxia). The data obtained could help to increase the awareness of the possibilities of SpO2 monitoring using smartwatches in medical conditions that are manifested by a decrease in SpO2 level over a longer time period, where measurement with a conventional oximeter is impractical.

ELIGIBILITY:
Inclusion Criteria:

* Passing the initial examination, which will determine the following data: wrist circumference, heart rate, blood pressure and blood oxygen saturation

Exclusion Criteria:

* pregnancy
* severe cardiovascular conditions
* severe asthma or other severe respiratory conditions
* injury to the upper limbs or hands that could affect the peripheral perfusion
* diabetes
* hypotension or hypertension

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-28 (Estimated)

PRIMARY OUTCOMES:
Similarity of SpO2 readings | Under 1 hour
  The agreement of SpO2 measurements of every model of smartwatches and reference pulse oximeter will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Rafl, PhD., Principal Investigator — Czech Technical University in Prague
Locations (1):
- Czech Technical University in Prague, Kladno, Czechia

REFERENCES:
- [Background] Rafl J, Bachman TE, Rafl-Huttova V, Walzel S, Rozanek M. Commercial smartwatch with pulse oximeter detects short-time hypoxemia as well as standard medical-grade device: Validation study. Digit Health. 2022 Oct 11;8:20552076221132127. doi: 10.1177/20552076221132127. eCollection 2022 Jan-Dec. PMID 36249475